CLINICAL TRIAL: NCT06395883
Title: Dynamics in Bone Turnover Markers During and After Short-term Glucocorticoid Treatment in Patients With an Inflammatory Joint Disease - the BOOGIE Study
Brief Title: Dynamics in Bone Turnover Markers During and After Short-term Glucocorticoid Treatment in Patients With an Inflammatory Joint Disease
Acronym: BOOGIE
Status: Recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other)
Responsible Party: Sponsor
Other Study IDs: DS-00846
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis; Osteoporosis, Steroid Induced; Inflammatory Rheumatism
Keywords: Bone turnover; Bone turnover markers; Glucocorticoids
MeSH Terms: conditions — Osteoporosis; Rheumatic Fever | interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- RApre: Patients with a new diagnosis of rheumatoid arthritis and indication for initiating DMARD treatment with a bridging of oral glucocorticoid treatment. Women should be premenopausal and men younger than 50 years.
  Interventions: Drug: Glucocorticoid Effect
- RApost: Patients with a new diagnosis of rheumatoid arthritis and indication for initiating DMARD treatment with a bridging of oral glucocorticoid treatment. Women should be postmenopausal and men older than 50 years.
  Interventions: Drug: Glucocorticoid Effect
- SpA: Patients with a new diagnosis of spondyloarthritis and indication of DMARD treatment without glucocorticoid treatment. Women should be premenopausal and men younger than 50 years.
- PsA: Patients with a new diagnosis of psoriatic arthritis and indication of DMARD treatment without glucocorticoid treatment. Women should be premenopausal and men younger than 50 years.
- IA: Patients with an inflammatory joint disease on stable DMARD treatment weith indication of intraarticular glucocorticoid injection. Women should be premenopausal and men younger than 50 years.
  Interventions: Drug: Glucocorticoid Effect
- IM: Patients with an inflammatory joint disease on stable DMARD treatment weith indication of intramuscular glucocorticoid injection. Women should be premenopausal and men younger than 50 years.
  Interventions: Drug: Glucocorticoid Effect

INTERVENTIONS:
Drug: Glucocorticoid Effect — Patients with or without glucocorticoid treatment will be observed regarding the level of bone turnover markers (P1NP and CTX1) every 4 weeks til 6 months after the last glucocorticoid dose.
  Groups: IA; IM; RApost; RApre

SUMMARY:
Bone turnover markers (BTMs) are recommended as an important tool in follow-up of osteoporosis treatment. However, there is a lack of knowledge in the reliability of BTMs during and after glucocorticoid treatment. Glucocorticoids suppresses BTMs during treatment with at least 30% and, moreover, glucocorticoids increase the risk of fractures. Patients with an inflammatory joint disease are at increased risk of osteoporosis, and disease flares are often treated with glucocorticoids, which in turn can lead to loss in reliability of the BTMs in patients who also are on osteoporosis treatment.

There is a need of more knowledge on BTM changes during and after glucocorticoid treatment for optimized patientcare, reduced risk of side effects and reduced health economic costs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of inflammatory rheumatic joint disease
* indication of disease modifying treatment initiation with or without glucocorticoids OR
* stable DMARD treatment with parenteral glucocorticoid injection

Exclusion Criteria:

* known osteoporosis or osteoporosis treatment
* women during the transitory phase
* oestrogen treatment
* any fracture within the last year
* chronic glucocorticoid treatment
* glucocorticoid treatment within the last year prior to inclusion
* active cancer
* kidney failure

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of rheumatoid arthritis or spondyloarthritis or psoriatic arthritis
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
P1NP level 3 months after glucocorticoid termination | september 2024 til december 2025
  P1NP in a blood sample

SECONDARY OUTCOMES:
P1NP level 6 months after glucocorticoid termination | september 2024 til december 2025
  P1NP in a blood sample
CTX1 level 3 and 6 months after glucocorticoid termination | september 2024 til december 2025
  CTX1 in a blood sample
P1NP and CTX1 dynamic until 6 months after treatment of inflammation without glucocorticoids | september 2024 til december 2025
  P1NP and CTX1 in a blood sample

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Vestre Viken HF, Drammen, Drammen
  - Diakonhjemmet hospital, Oslo

IPD SHARING:
Plan to Share IPD: No